CLINICAL TRIAL: NCT06377852
Title: Comparing Oral Drug Dosing Strategies in Older Patients With Metastatic Breast Cancer to Maximize Tolerance and Reduce Discontinuation: The CDK4/6 Inhibitor Dosing Knowledge (CDK) Study
Brief Title: The CDK4/6 Inhibitor Dosing Knowledge (CDK) Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: American Society of Clinical Oncology (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00075309
Record Dates: First submitted 2024-04-08; First posted 2024-04-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; ribociclib

STUDY DESIGN:
Intervention Model Description: 500 patients will be enrolled, 250 per arm (Arm 1 being indicated dose, Arm 2 being titrated dose).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Indicated Dose (Experimental): Arm 1 of the study is the indicated dosing regimen, provided in the FDA approved drug label: participants will start cycle 1 with either 125mg dose of palbociclib or 600mg dose of ribociclib, in combination with endocrine therapy (AI or fulvestrant).
  Interventions: Drug: Palbociclib 125mg; Drug: Ribociclib 600mg
- Arm 2: Titrated Dose (Experimental): Arm 2 is the titrated dosing regimen: participants will start cycle 1 with either 100 mg or 75 mg dose of palbociclib or 400 mg or 200 mg dose of ribociclib, in combination with endocrine therapy (AI or fulvestrant). For cycle 2 and for subsequent cycles, escalation to the indicated dose will be based on treatment tolerance.
  Interventions: Drug: Ribociclib; Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib 125mg — Arm 1: Indicated dosing for palbociclib (125 mg orally daily on days 1-21 of 28-day cycle)
  Arms: Arm 1: Indicated Dose
Drug: Ribociclib 600mg — Arm 1: Indicated dosing of ribociclib (600 mg orally daily on days 1-21 of 28-day cycle)
  Arms: Arm 1: Indicated Dose
Drug: Ribociclib — Arm 2: Titrated dosing approach with the same schedule but starting at a lower dose of ribociclib (400 mg or 200 mg) and escalating the dose if well-tolerated in combination with provider/patient choice of endocrine therapy.
  Arms: Arm 2: Titrated Dose
Drug: Palbociclib — Arm 2: Titrated dosing approach with the same schedule but starting at a lower dose of palbociclib (100 mg or 75 mg) and escalating the dose if well-tolerated in combination with provider/patient choice of endocrine therapy.
  Arms: Arm 2: Titrated Dose

SUMMARY:
The purpose of this study is to generate evidence on an alternative dosing strategy for CDK4/6 inhibitors to help more patients with Metastatic Breast Cancer (MBC) (age ≥ 65 years) tolerate side effects and stay on treatment longer, to derive the most clinical benefit from these drugs.

The primary objective of the CDK Study is to compare time to treatment discontinuation (TTD) on the approved dosing for palbociclib (125 mg orally daily on days 1-21 of 28-day cycle) or ribociclib (600 mg orally daily on days 1-21 of 28-day cycle) vs. TTD using titrated dosing approach with the same schedule but starting at a lower dose of palbociclib (100 mg or 75 mg) or ribociclib (400 mg or 200 mg) and escalating the dose if well-tolerated in combination with provider/patient choice endocrine therapy (aromatase inhibitor (AI) or fulvestrant) in patients age 65 or older with HR+/HER2- MBC. The secondary and exploratory objectives will generate evidence needed to personalize treatment decisions by comparing patient-centric secondary outcomes and evaluating baseline factors.

Together with their treating physician, participants will choose the CDK4/6 inhibitor (palbociclib or ribociclib) and which endocrine therapy (aromatase inhibitor or fulvestrant) of their choice but will be randomized to either Arm 1 (indicated dosing) or Arm 2 (titrated dosing).

Note: Telehealth visits are allowed at any time per institutional guidelines. In addition, the study allows for remote consenting per institutional guidelines.

DETAILED DESCRIPTION:
The CDK4/6 Inhibitor Dosing Knowledge Study (CDK Study) will study CDK4/6 inhibitor dosing regimens in patients 65 or older with Metastatic Breast Cancer (MBC). The overarching goal of this pragmatic, randomized trial is to compare an "indicated" dosing approach, as listed on the FDA-approved drug label, that starts at the full dose of a CDK4/6 inhibitor (palbociclib or ribociclib) with dose reduction based on tolerability versus a "titrated" dosing approach that starts at a lower dose of a CDK4/6 inhibitor and then titrates up to full dose as tolerated. CDK4/6 inhibitors will be given in combination with endocrine therapy (either an aromatase inhibitor (AI) or fulvestrant) based on the choice of the treating clinician.

The primary endpoint will be time to treatment discontinuation (TTD), defined as the time from randomization to last dose of the CDK4/6 inhibitor. The hypothesis is that starting low and escalating as tolerated will help older patients (> 65 years) stay on therapy longer. Eligibility criteria are broad to allow patients who are not typically included in clinical trials to participate, allowing for a more representative sample of participants. The investigators will conduct sub-group analyses based on age (65-74 years vs. ≥75 years) and baseline frailty scores. This study builds upon the lessons learned from prior studies with CDK4/6 inhibitors. The investigators will augment the standard assessment of treatment toxicities assessed by the health care team with prospectively collected patient-reported outcomes data to better reflect how participants tolerate the different dosing approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Hormone receptor positive (HR+) HER2 negative metastatic breast cancer. Cut-off values for positive/negative staining should be as per standard practice in accordance with ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines. Verification of histology is preferred at the time of recurrence and where not possible or necessary in the judgment of the treating physician, the study will accept histology from the initial diagnosis.
2. Candidate for planned endocrine therapy in combination with 1st use of palbociclib or ribociclib, in the metastatic setting. The planned endocrine partner can be an aromatase inhibitor (letrozole, anastrozole, exemestane) or fulvestrant, selected through patient/provider choice.
3. Aged 65 years or older
4. Adequate bone marrow and organ function. Laboratory values must be within normal institutional limits, or within ranges as indicated below, or demonstrate minor abnormalities that are deemed clinically non-significant by the investigator.

   * Absolute neutrophil count ≥ 1,000/µL
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (participants with documented Gilbert's disease are allowed total bilirubin up to 5X ULN)
   * AST (SGOT)/ALT (SGPT) <3 x institutional ULN, or ≤ 5 x ULN for subjects with documented metastatic disease to the liver.
5. Baseline QTc ≤ 480 ms (only for ribociclib patients)
6. Ability to understand and the willingness to provide informed consent. Note: Remote consent is allowed per institutional guidelines.

Exclusion Criteria:

1. Previous treatment with a CDK4/6 inhibitor for metastatic breast cancer, or previous treatment within the past 12 months with a CDK4/6 inhibitor in the neo/adjuvant breast cancer setting.
2. Received greater than 30 days (in the metastatic setting) of the specific endocrine therapy agent planned as partner to the CDK4/6 inhibitor in the study at the time of randomization.
3. Known history of intolerance or allergy to the planned agents used in this trial.
4. Uncontrolled intercurrent illness that, as evaluated by the treating clinician, would hinder compliance with study requirements.
5. Concurrent therapy with other investigational agents.
6. Rapidly progressive brain metastases.
7. Active or chronic Hepatitis B or C are eligible provided they meet liver function laboratory criteria and are not on medication with a known interaction with the study agents.
8. Current use of drugs that have known potential to prolong the QT interval (e.g., antiarrhythmic drugs), for patients on ribociclib. Note: If concomitant use cannot be avoided, monitor ECG when initiating, during concomitant use, and as clinically indicated. Refer to crediblemeds.org as a resource.
9. Prior or concurrent malignancies that are undergoing active treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to Treatment Discontinuation (TTD) | up to 48 months
  Our primary outcome is time to CDK4/6 inhibitor discontinuation (TTD): the number of days between randomization and the last day the patient takes any dose of the same CDK4/6 inhibitor (regardless of drug holds, dose changes

SECONDARY OUTCOMES:
Toxicity (grade 3-4 AEs) | up to 48 months
  Assessed in each arm of the study and study drug
Event-Free survival (EFS) | up to 48 months
  Assessed in each arm of the study and study drug
Quality of life assessed by patient reported outcomes | up to 48 months
  PROMIS-29 (3 domains of 12 questions, physical function, fatigue, participation in social activities), FACT-G Item GP5 (1 question)
Time to dose reduction and escalation | up to 48 months
  For titrated arm. Assessed in each arm of the study and study drug
Reason for not escalating | up to 48 months
  Assessed in each arm of the study and study drug
Treatment received (missed doses, cumulative dose, etc.) | up to 48 months
  Assessed in each arm of the study and study drug
Healthcare utilization (ED visits, hospital admissions, etc.) | up to 48 months
  ED visits, hospital admissions, etc., assessed in each arm of the study and study drug
Body Mass Index | up to 48 months
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gralow, MD, Principal Investigator — American Society of Clinical Oncology
Locations (60):
- United States (60):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Cherry Creek Medical Center, Denver, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Smilow Cancer Hospital Care Center - Derby, Derby, Connecticut
  - Smilow Cancer Hospital Care Center - Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center - Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital at Saint Francis, Hartford, Connecticut
  - Yale University/Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center - North Haven, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center - Torrington, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center - Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterbury, Waterbury, Connecticut
  - Smilow Cancer Hospital - Waterford, Waterford, Connecticut
  - Miami Cancer Institute, Miami, Florida
  - Miami Cancer Institute, Plantation, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion, Savannah, Georgia
  - The University of Kansas Cancer Center, Westwood, Kansas
  - The Jackson Laboratory (JAX) - Harold Alfond Center for Cancer Care, Augusta, Maine
  - The Jackson Laboratory (JAX) - Northern Light Cancer Care, Brewer, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Brigham Cancer Center Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Brigham Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber Brigham Cancer Center at South Shore Health, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - Penn Medicine - Princeton Health, Plainsboro, New Jersey
  - Lovelace Medical Center - Saint Joseph Square, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - The University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Levine Cancer Institute, Albemarle, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute, Concord, North Carolina
  - Levine Cancer Institute, Forest City, North Carolina
  - Levine Cancer Institute, Gastonia, North Carolina
  - Levine Cancer Institute, Huntersville, North Carolina
  - Levine Cancer Institute, Lincolnton, North Carolina
  - Levine Cancer Institute, Matthews, North Carolina
  - Levine Cancer Institute, Monroe, North Carolina
  - Levine Cancer Institute, Shelby, North Carolina
  - Penn Medicine - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Medicine - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Penn Medicine - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Penn Medicine - Chester County Hospital, West Chester, Pennsylvania
  - Smilow Cancer Hospital - Westerly, Westerly, Rhode Island
  - St. Joseph's Candler Bluffton Campus, Bluffton, South Carolina
  - SC Cancer Specialists - Hilton Head at St. Joseph's/Candler, Hilton Head Island, South Carolina
  - Levine Cancer Institute, Rock Hill, South Carolina
  - Baptist Memorial Healthcare, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No